CLINICAL TRIAL: NCT05306275
Title: A Phase 1, Randomized, Open-label, Parallel-group Study to Compare the Pharmacokinetic Properties of CSL312 Administered by Subcutaneous Prefilled Syringe Assembled to Autoinjector to Prefilled Syringe Assembled to Needle Safety Device in Healthy Adult Subjects
Brief Title: A Study to Compare the Pharmacokinetics of CSL312 Administered by Prefilled Syringe Assembled to Autoinjector to the Pharmacokinetics Administered by Prefilled Syringe Assembled to Needle Safety Device in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CSL312_1004
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- CSL312 AI Abdomen (Experimental): CSL312 administered subcutaneously (SC) in the abdomen via a prefilled syringe assembled to an autoinjector (AI)
  Interventions: Drug: CSL312
- CSL312 AI Thigh (Experimental): CSL312 administered SC in the thigh via a prefilled syringe assembled to an AI
  Interventions: Drug: CSL312
- CSL312 AI Arm (Experimental): CSL312 administered SC in the upper arm via a prefilled syringe assembled to an AI
  Interventions: Drug: CSL312
- CSL312 NSD Abdomen (Experimental): CSL312 administered SC in the abdomen via a prefilled syringe assembled to a needle safety device (NSD)
  Interventions: Drug: CSL312
- CSL312 NSD Thigh (Experimental): CSL312 administered SC in the thigh via a prefilled syringe assembled to a NSD
  Interventions: Drug: CSL312
- CSL312 NSD Arm (Experimental): CSL312 administered SC in the upper arm via a prefilled syringe assembled to a NSD
  Interventions: Drug: CSL312

INTERVENTIONS:
Drug: CSL312 — Factor XIIa antagonist monoclonal antibody for subcutaneous use
  Other Names: Gardacimab

SUMMARY:
This is an open-label, parallel-group, phase 1, single center study to assess the relative bioavailability of CSL312 administered subcutaneously via a prefilled syringe assembled to an autoinjector compared to a prefilled syringe assembled to a needle safety device in healthy, adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male or female 18 to 55 years of age
* Body weight in the range of ≥ 50 kg and ≤ 100 kg, with a body mass index (BMI) of ≥ 18 kg/m2 and ≤ 30 kg/m2

Exclusion Criteria:

* Received any live viral or bacterial vaccinations within 8 weeks of Screening or is expected to receive any live virus or bacterial vaccinations during the study or up to 4 months after last administration of the investigational product.
* Evidence of current active infection, including severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2).
* Blood pressure or pulse rate measurements outside the normal range for the subject's age

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of CSL312 | Up to 85 days post-dose
Area under the concentration-time curve (AUC) from time 0 extrapolated to infinite time (AUC0-inf) of CSL312 | Up to 85 days post-dose

SECONDARY OUTCOMES:
Number and percentage of subjects experiencing adverse events (AEs) | Up to 85 days post-dose
Number and percentage of subjects experiencing serious adverse events (SAEs) | Up to 85 days post-dose
Number and percentage of subjects experiencing adverse events of special interest (AESIs) | Up to 85 days post-dose
Number and percentage of subjects developing Anti-CSL312 antibodies | Up to 85 days post-dose
Number and percentage of subjects with clinically significant laboratory abnormalities that are reported as AEs | Up to 85 days post-dose
Number and percentage of subjects with injection site reactions by severity | Up to 48 hours post-injection
Time to maximum plasma concentration (Tmax) of CSL312 | Up to 85 days post-dose
AUC from time 0 to the last measurable concentration (AUC0-last) of CSL312 | Up to 85 days post-dose
Half-life (t1/2) of CSL312 | Up to 85 days post-dose
Apparent clearance (CL/F) of CSL312 | Up to 85 days post-dose
Apparent volume of distribution (Vz/F) of CSL312 | Up to 85 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (1):
- Anaheim Clinical Trials, LLC, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (ie FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.